CLINICAL TRIAL: NCT03687112
Title: National Bank Alzheimer
Acronym: BNA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 18-DSP-03
Record Dates: First submitted 2018-09-20; First posted 2018-09-27 (Actual); Last update posted 2018-09-27 (Actual); Status verified 2018-09

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Alzheimer desease and related disorders: Alzheimer desease and related disorders
  Interventions: Other: non ontervention / observational study

INTERVENTIONS:
Other: non ontervention / observational study — non intervention

SUMMARY:
The Alzheimer's disease (MY) is a major problem of public health. The French National Database Alzheimer ( BNA) registers(records) all the medical acts made by units of memory(report) and of independent specialists in France.

In 2008, the national Plan Alzheimer 2008 - 2012 had for objective to strengthen the search(research) on the Alzheimer's disease (MY) and for related disorders(confusions), to promote an early diagnosis and to improve at the same time the management of the patients and to support careers(quarries). A specific part(party) of this plan gave rise to the creation of the French national database Alzheimer ( BNA) to supply epidemiological data as well as indicators of activity. Since 2009 The information collected(taken in) in the BNA consists of a set(group) limited by data (CIMA of information minimum Corpus Alzheimer) concerning the demographic, clinical and diagnostic data defined by national consensus. The number of variables is limited to facilitate and to improve the participation in this national database. The participants are the Centers Report (CM)((LECTURE)) and Center Memory(Report) of Resources and Search(Research) (CMRR) and independent specialists. In 2015 more than 500 Centers send CIMA to the BNA.

The plan Disease Neurodegenerative 2014 - 2019 wishes to pursue and to amplify the BNA.

ELIGIBILITY:
Inclusion Criteria:

* patients consulting in French Memory Centres

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Alzheimer desease and related disorders patients
Sampling Method: Non-Probability Sample
Dates: Start 2009-01-01 (Actual); Primary Completion 2009-01-01 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Evolution of the morbi-mortality | 16 years
  number of people suffering from a disease
Evolution of the morbi-mortality | 16 years
  number of deaths

SECONDARY OUTCOMES:
number of the miscellaneous determiners of Access to healthcare or diagnosis | 16 years
  number of the determiners of the access to healthcare and diagnosis

OTHER OUTCOMES:
New therapeutic plans | 16 years
  Participate in the evaluation of new therapeutic plans of care

CONTACTS AND LOCATIONS:
Locations (1):
- Nice University Hospital, Nice, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mouton A, Plonka A, Fabre R, Tran TM, Robert P, Macoir J, Manera V, Gros A. The course of primary progressive aphasia diagnosis: a cross-sectional study. Alzheimers Res Ther. 2022 May 10;14(1):64. doi: 10.1186/s13195-022-01007-6. PMID 35538502